CLINICAL TRIAL: NCT00228943
Title: The Role of Serotonin in Hot Flashes After Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: Janet Carpenter, PhD, RN, Indiana University School of Nursing
Organization: Indiana University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 0501-03; DOD-BC043199; 043199
Record Dates: First submitted 2005-09-14; First posted 2005-09-29 (Estimated); Results first posted 2008-12-10 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer survivorship; Hot Flashes; Serotonin
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute tryptophan depletion (Experimental): Full-strength tryptophan depletion
  Interventions: Dietary Supplement: Acute tryptophan depletion
- Control (Active Comparator): Half-strength tryptophan depletion drink used as a control
  Interventions: Dietary Supplement: Half-strength tryptophan depletion (Control)

INTERVENTIONS:
Dietary Supplement: Acute tryptophan depletion — L-alanine (5.5g), L-arginine (4.9g), L-cysteine (2.7g), glycine (3.2g), L-histidine (3.2g), L-isoleucine (8.0g), L-leucine (13.5g), L-lysine (11.0g), L-methionine (3.0g), L-phenylalanine (5.7g), L-proline (12.2g), L-serine (6.9g), L-threonine (6.9g), L-tyrosine (6.9g), L-valine (8.9g)
  Arms: Acute tryptophan depletion
Dietary Supplement: Half-strength tryptophan depletion (Control) — L-alanine (1.4g), L-arginine (1.2g), L-cysteine (0.7g), glycine (0.8g), L-histidine (0.8g), L-isoleucine (2.0g), L-leucine (3.4g), L-lysine (2.8g), L-methionine (0.8g), L-phenylalanine (1.4g), L-proline (3.1g), L-serine (1.7g), L-threonine (1.7g), L-tyrosine (1.7g), L-valine (2.2g), and fillers (7.95g).
  Arms: Control

SUMMARY:
The purpose of this proposal is to improve our understanding of the role of tryptophan and serotonin in hot flashes. The main hypothesis is that alterations in tryptophan and serotonin levels are involved in the induction of hot flashes in women with breast cancer and genetic variations in the serotonin receptors and transporters also play a role.

DETAILED DESCRIPTION:
Among women with breast cancer, hot flashes are a frequent, severe and bothersome symptom. For this group, hot flashes are negatively related to mood, affect, and daily activities and can compromise compliance with life-saving medications (e.g., tamoxifen). Over 60% of breast cancer survivors report hot flashes, with 59% stating they are extremely severe and 44% reporting them to be extremely bothersome. Unfortunately, limitations in our understanding of hot flash physiology limit clinicians' abilities to fully treat this symptom. Although the current non-hormonal treatment of choice for hot flashes after breast cancer targets the central serotonin system (e.g., paroxetine, venlafaxine), the role of serotonin in hot flashes has not been directly tested. Because the effectiveness of these agents has been based largely on improvement in subjective reporting of hot flashes, it is not clear whether benefits are due to physiological effects on hot flashes or due to improvements in mood or other related symptoms. In addition, these and other currently available treatments are not acceptable, appropriate, or effective for all women with breast cancer. Understanding the physiological mechanisms involved in hot flashes after breast cancer will enable us to develop more targeted behavioral and/or pharmacological therapies to be used in lieu of, or in addition to, currently available therapies so that we can eradicate hot flashes and improve the quality of life for women with breast cancer.

Results implicating direct effects of tryptophan and serotonin on objective hot flashes will help guide the development of improved interventions for alleviating hot flashes in women with breast cancer. These interventions may target the central serotonin system either behaviorally (e.g., diet) or pharmacologically (e.g., alternative drug therapeutics). If direct manipulation of tryptophan and serotonin does not affect hot flashes, these findings will be equally as useful in guiding future research on non-serotonin related etiologies and interventions. Findings from this study will ultimately be used to eradicate hot flashes as a frequent, severe and bothersome breast cancer treatment related condition, thereby, improving quality of life for all women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willing and able to provide informed consent
* Reporting daily hot flashes
* Able to read, write, and speak English
* Postmenopausal to limit sample variability (> 12 months amenorrhea)
* Greater then 1 month but < 5 years post-treatment (surgery, radiation, chemotherapy) for non-metastatic breast cancer.
* These criteria allow inclusion of women successfully treated for recurrent breast cancer since there is no known reason to exclude them. Menopausal status is assessed using self-reports due to problems in reliably measuring follicle-stimulating hormone levels and estradiol in tamoxifen users.

Exclusion Criteria:

* Exclusion criteria are current depression, history of migraines or hepatitis, abnormal chemistry profile (e.g., sodium, potassium, glucose), or a positive urine drug screen for illegal substances.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-07; Primary Completion 2007-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet S Carpenter, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Carpenter JS, Yu M, Wu J, Von Ah D, Milata J, Otte JL, Johns S, Schneider B, Storniolo AM, Salomon R, Desta Z, Cao D, Jin Y, Philips S, Skaar TC. Evaluating the role of serotonin in hot flashes after breast cancer using acute tryptophan depletion. Menopause. 2009 Jul-Aug;16(4):644-52. doi: 10.1097/gme.0b013e318199e9f6. PMID 19265726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a Midwestern outpatient cancer clinic from 2005 to 2007.
Pre-assignment Details: 260 women were screened, 39 of whom were not interested, 162 were found ineligible.
Groups:
- Full Strength Acute Tryptophan Depletion and Control: Subjects were randomized to receive both a full-strength acute tryptophan depletion drink and half-strength tryptophan depletion drink (control). Some participants received the full-strength drink first for week 1 and then crossed-over to the half-strength (control) drink for week 2; the other participants received the half-strength (control) drink for week 1 and then crossed over to the full-strength drink for week 2.
Period: Week 1
Arm/Group | Full Strength Acute Tryptophan Depletion and Control
Started | 28
Completed | 28
Not Completed | 0
Period: Week 2
Arm/Group | Full Strength Acute Tryptophan Depletion and Control
Started | 28
Completed | 27
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Sample: Consented subjects in the entire sample were randomized to one of two groups for the cross-over design study. One group of subjects received a full-strength tryptophan depletion drink during week 1 followed by a half-strength (control) drink week 2. The other group of subjects received a half-strength tryptophan depletion (control) drink during week 1 followed by a full-strength drink week 2.
  The final analysis combined groups to compare full strength versus control.
Arm/Group | Entire Sample
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Serum Tryptophan Levels
Description: Mean serum tryptophan levels (blood draw) at the end of the nadir period.
Time Frame: baseline, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours
Population: The number of subjects with complete serum data for both arms of the study were analyzed.
Measure: Mean (Standard Deviation); unit: nmol/ml
Arm/Group | Full Strength Acute Tryptophan Depletion | Half-Strength Tryptophan Depletion - Control
Number analyzed (Participants) | 24 | 23
nmol/ml | 0.0034 (.0027) | 0.02 (0.02)

2. Primary Outcome: Objective Subject Hot Flash Frequency
Description: Mean of the 24 hour monitoring sessions for each patient based on one 24 hour monitoring session after each intervention using an electronic monitor.
Time Frame: One 24 hour monitoring session per week for 8 weeks
Population: Subjects with completed hot flash data during both arms of study.
Measure: Mean (Standard Deviation); unit: frequency of hot flashes
Arm/Group | Full Strength Acute Tryptophan Depletion | Half-Strength Tryptophan Depletion - Control
Number analyzed (Participants) | 27 | 27
frequency of hot flashes | 2.30 (2.92) | 2.62 (3.29)

ADVERSE EVENTS:
Groups:
- Full Strength Acute Tryptophan Depletion; Half-Strength Tryptophan Depletion - Control: No adverse events
Arm/Group | Full Strength Acute Tryptophan Depletion | Half-Strength Tryptophan Depletion - Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No